CLINICAL TRIAL: NCT01171573
Title: Identification of Disease Susceptibility Genes Associated With Development and Clinical Characteristics of Primary Inflammatory Muscle Diseases, PM, DM and IBM.
Brief Title: Investigating Genes in Patients With Polymyositis and Dermatomyositis
Acronym: UKMYONET
Status: Active, not recruiting | Type: Observational
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Hector Chinoy, Senior Lecturer/Consultant Rheumatologist, University of Manchester
Other Study IDs: Ollier-002
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Myositis
Keywords: Polymyositis; Dermatomyositis; Inclusion Body Myositis
MeSH Terms: conditions — Myositis; Polymyositis; Dermatomyositis; Myositis, Inclusion Body | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Myositis Patients: Cases with myositis PM DM IBM Venepuncture
  Interventions: Procedure: Venepuncture
- Healthy controls: Control
  Interventions: Procedure: Venepuncture

INTERVENTIONS:
Procedure: Venepuncture — Venepuncture - Taking blood

SUMMARY:
Polymyositis (PM), dermatomyositis (DM) and inclusion body myositis (IBM)belong to a group of inflammatory muscle disorders, of unknown cause, that are characterised by skeletal muscle inflammation and progressive muscular weakness, which can be debilitating and chronic in nature (occasionally fatal).

The current treatment options for these conditions are steroids and various other immunosuppressive drugs. However, these are usually only partially effective at reducing symptoms, and their toxic side effects also limit their usefulness. In order to develop more specific treatments for myositis in the future (and therefore more effective), it is important to understand the exact mechanisms that cause the disease in the first instance. In other similar inflammatory diseases such as rheumatoid arthritis (RA) and systemic lupus (SLE), it is known that changes to the Human Leukocyte Antigen(HLA), as well as certain inflammatory cytokines, are involved in both the development and expression of the disease.

As many of the inflammatory mechanisms that cause damage in PM, DM and IBM are similar to those in RA and SLE, it seems likely that similar genetic factors will also be involved in the development and expression of PM, DM and IBM.

In order to understand the genetic aspects / causes of myositis, and ultimately develop more effective treatment therapies in the future, patients with PM, DM or IBM, will be asked to give 20 mls of blood. These blood samples, along with the patient's clinical details, will then be sent to the Centre for Integrated Genomic Medical Research (CIGMR), at The University of Manchester, where all of the genetic analyses will take place. By understanding the genetic cause of the disease, it should be possible to design specific drugs for treating the condition in the future.

DETAILED DESCRIPTION:
In order to understand the genetic aspects / causes of myositis, and ultimately develop more effective treatment therapies, it will be necessary to collect blood samples and clinical details from around 1000 patients with myositis. As the condition is very rare, it will not be possible to get the required number of patients from one centre alone, and therefore, a collaborative, multicentred approach will be needed. Consultant rheumatologists and neurologists throughout the UK, who have patients with PM, DM or IBM, will be approached, and asked if they would like to officially enter into the myositis genomic multicentred study. Once ethical and R&D approval has been granted, consultants will be named as the 'Principal Investigators' at each of these 'research sites' and could then start to recruit suitable patients into the study.

Patients from each research site, with definite PM, DM or IBM, will be asked by their own consultants (Principal Investigator) to give 20 mls of blood via venepuncture for genetic and antibody analysis. The PI will also complete a clinical/laboratory proforma, for each patient, regarding their disease characteristics, to allow subsequent confirmation that patients' disease is indeed definite, and this proforma and the blood sample will be sent to CIGMR. All of the genetic analyses, will take place at CIGMR, but storage of clinical details and certain patient identifiers will be stored at SRFT on a password protected NHS tust computer.

This study will be co-ordinated by Dr RG Cooper through the Rheumatic Diseases Centre, Salford Royal NHS Foundation Trust (SRFT), and Professor Bill Ollier from the Centre for Integrated Genomic Medical Research unit (CIGMR), Stopford Building, Manchester University.

ELIGIBILITY:
Inclusion Criteria:

Cases must fulfil Bohan and Peter Diagnostic Criteria for Adult PM/DM

1. Symmetrical weakness of limb-girdle muscles and/or anterior neck flexors.
2. Muscle biopsy evidence typical of myositis.
3. Elevation of serum skeletal muscle enzymes.
4. Typical EMG features of myositis.
5. Typical DM rash, including:

Probable / definite PM: at least 3 of items 1-4 +ive. Probable / definite DM: item 5 & at least 2 of items 1-4 +ive.

Exclusion Criteria:

* Patients below the age of 18 years
* Patients with myositis secondary to alcohol or drug abuse, non abusive drug ingestion (e.g with statins, fibrates etc)
* Patients with myositis following a recent viral illnesses.
* Patients unable to consent for themselves due to diminished mental capacity
* Patients that can not speak sufficiently good English.
* Patients unwilling to give blood sample.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified at their routine attendance of myositis clinics at participating centres, by the study PI. Before recruitment, each prospective candidate will be given a full explanation of the study, provided with a patient information sheet (PIS) and consent form to read, and given the opportunity to ask any questions that may arise. Once all questions have been answered and the Principal Investigator is assured that the individual understands what is required, informed consent can then be sought.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To identify any disease susceptibility genes associated with development and clinical characteristics of primary inflammatory muscle diseases, PM, DM and IBM. | 20 years
  Blood sample, DNA analysis, along with clinical data, matching genotype with phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dr Cooper, Principal Investigator — SRFT
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom